CLINICAL TRIAL: NCT07233473
Title: Prospective, Multicentric, Single Arm Clinical Investigation to Assess the Effectiveness and Safety of Multi-Gyn UT Protect Gel for Prevention of Recurrent Urinary Tract Infections
Brief Title: Evaluation of the Effectiveness and Safety of a Vaginal Gel for Prevention of Recurrent Urinary Tract Infections
Acronym: UTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-1775-U5
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Urinary Tract Infections (UTIs)
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Vaginal gel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study product (Experimental): Multi-Gyn UT Protect gel
  Interventions: Device: Multi-Gyn UT Protect gel

INTERVENTIONS:
Device: Multi-Gyn UT Protect gel — Vaginal gel

SUMMARY:
Urinary Tract Infections (UTIs) are among the most common bacterial infections. Although they are typically treated effectively with antibiotics, recurrence is a frequent and troublesome issue.

This clinical trial aims to evaluate the safety and effectiveness of Multi-Gyn UT Protect gel in preventing the recurrence of UTIs. The trial will involve 50 adult female participants who have experienced a UTI in recent months but do not currently have an active infection.

Each participant will apply the gel twice a week for four months. They will be monitored throughout this period to assess whether participants develop the reappearance of UTI symptoms.

The primary objective is to determine how many participants do not experience a recurrence of UTI by the end of the four-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 84 years old.
2. Sex: Female.
3. Subject suffering from uncomplicated recurrent urinary tract infections: ≥ 4. UTIs within 12 months or ≥ 2 within 6 months.
4. Subject having given freely and expressly her informed consent.
5. Subject using a contraceptive regimen recognized as effective (pill, implant, Intra Uterine Device (IUD), condoms) since at least 12 weeks before inclusion visit and during the whole study. If subject use condoms as contraceptive regimen, a delay of 6 hours between application and sexual intercourse must be respected.
6. Subject affiliated to a health social security system.
7. Subject cooperative and aware of the device's modalities of use and the necessity and duration of the follow-up visits so that perfect adhesion to the protocol can be expected.

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who gave birth in the 3 previous months.
3. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
4. Subject in a social or sanitary establishment.
5. Subject suspected to be non-compliant according to the investigator's judgment.
6. Subject having received 6000 euros indemnities for participation in clinical research in the 12 previous months, including participation in the present study.
7. Subject enrolled in another clinical trial or which exclusion period is not over.
8. Subject with history of complicated urinary tract infection.
9. Subject with urinary tract infection at the time of inclusion.
10. Subject with vaginal mycosis infection in the last 3 weeks.
11. Subject with recurrent vaginal mycosis (more than 2 in the last 6 months).
12. Subject having a known allergy or hypersensitivity to one of the components of the investigational device.
13. Subject suffering from a sexually transmitted gynaecological infection or aerobic vaginitis (including gonorrhoea, chlamydia trachomatis or mycoplasma genitalium infection with cervicitis, urethritis, salpingitis).
14. Subject with history of hormone-dependent cancer or bladder cancer.
15. Subject with current genital malignancies.
16. Subject who had a chemotherapy treatment for a cancer in the 12 months before inclusion.
17. Subject who had a radiotherapy treatment in the genito-urinary area in the 12 months before inclusion.
18. Subject using treatment for urinary tract infection, vaginal conditions, vaginal infections, or other intravaginal treatment at the time of inclusion.
19. Subject using food supplements for prevention of urinary tract infection in the last 3 months.
20. Subject using antibiotics, corticoids or antifungal treatment for any reason in the 3 weeks before inclusion.
21. Subject using vaginal douches and who do not wish to refrain using them during the clinical investigation.
22. Subject with a pessary.
23. Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk.

Ages: 18 Years to 84 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women only
Enrollment: 50 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of Multi-Gyn UT Protect gel for the prevention of Urinary Tract Infection (UTI) relapse within 4 months | 4 months
  The number of patients without UTI relapse within 4 months will be summarized in frequency (N) and percentage (%), with a confidential interval CI 95%.

SECONDARY OUTCOMES:
To evaluate the effectiveness of Multi-Gyn UT Protect gel for the prevention of UTI relapse within 1, 2 and 3 months | 1, 2 and 3 months
  The number of patients without UTI relapse within 1, 2, 3 months will be summarized in frequency (N) and percentage (%), with a confidential interval CI 95% by time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No